CLINICAL TRIAL: NCT03047226
Title: Diagnosis of Lynch Syndrome Based on the Colorectal Core™ Platform in Colorectal Cancer Patients With the Loss of Staining by Immunohistochemistry (IHC) of Any of the Mismatch Repair (MMR) Proteins: An Open-label and Multi-center Study
Brief Title: Diagnosis of Lynch Syndrome Based on Next-generation Sequencing in Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Guangzhou Burning Rock Medical Examination Institute Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Ying Yuan, MD, Professor, Department of Medical Oncology, Second Affiliated Hospital, School of Medicine, Zhejiang University
Other Study IDs: RSKY2016019
Record Dates: First submitted 2017-01-23; First posted 2017-02-08 (Estimated); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Lynch Syndrome
Keywords: Lynch Syndrome; mismatch repair; microsatellite instability; next-generation sequencing; immunohistochemistry
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Microsatellite Instability | interventions — High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood, frozen tissue, paraffin tissue, Formalin-fixed tissue and RNA-later preserved tissue.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: next-generation sequencing — Use next-generation sequencing to test germline mutation and microsatellite instability.

SUMMARY:
The purpose of this study is to determine the proportion of patients diagnosed with Lynch syndrome in colorectal cancer patients with the loss of staining by immunohistochemistry (IHC) of any of the mismatch repair (MMR) proteins. Besides, this study aims to test the specificity and the sensitivity of detecting microsatellite instability (MSI) by next-generation sequencing, and to find out the consistency between IHC and MSI in colorectal cancer patients in China. In addition, researchers want to analyze the clinical characteristics and germline mutation of Lynch syndrome in Chinese population.

DETAILED DESCRIPTION:
1. Detect microsatellite instability (by next-generation sequencing and PCR capillary electrophoresis) and germline mutation (by next-generation sequencing) in probands.
2. Analyze the test outcome with clinical and family information to evaluate the germline mutation status preliminarily: likely pathogenic germline mutation, variant of uncertain significance, non-pathogenic germline mutation.
3. Verify the germline mutation in blood relatives whose proband has known likely pathogenic germline mutation or variant of uncertain significance.
4. Diagnose pathogenic germline mutation and non-pathogenic germline mutation based on clinical characteristics, family information and germline mutation test outcomes (including the outcomes of probands and blood relatives). Diagnose Lynch syndrome and the pathogenic germline mutation carriers in the included population.
5. Analyze the specificity and the sensitivity of detecting microsatellite instability (MSI) by next-generation sequencing; and analyze the consistency between IHC and MSI.
6. Analyze the clinical characteristics and germline mutation of Lynch syndrome in Chinese population.

ELIGIBILITY:
For probands, the inclusion criteria:

All of the following four points should be satisfied:

* Histological diagnosis of colorectal cancer;
* With the loss of staining by immunohistochemistry of any of the mismatch repair (MMR) proteins (MLH1, MSH2, MSH6, PMS2);
* With sufficient tumor tissue and normal tissue to test;
* Agree to provide basic information, clinical information and family history of cancer information.

For probands, the exclusion criteria:

* With at least one blood relative with known pathogenic germline mutation(s).

For blood relatives verifying germline mutation, the inclusion criteria:

All of the following three points should be satisfied:

* First- to second-degree blood relatives of probands with germline mutation(s).
* With Sufficient tumor tissue and normal tissue to test.
* Agree to provide basic information, clinical information and family history of cancer information.

For blood relatives verifying germline mutation, the exclusion criteria:

* Blood relatives who refuse to test.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The probands will be selected from colorectal cancer patients with the loss of staining by immunohistochemistry of any of the mismatch repair (MMR) proteins (MLH1, MSH2, MSH6, PMS2).
  The blood relatives verifying germline mutation will be selected from whose probands have germline mutation(s).
Sampling Method: Probability Sample
Enrollment: 311 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Pathogenic germline mutation | Upon completion of study, on average 2 years.
  Pathogenic germline mutation using next-generation sequencing with a targeted panel.

SECONDARY OUTCOMES:
Variant of uncertain significance of germline mutation | Upon completion of study, on average 2 years.
  Variant of uncertain significance of germline mutation using next-generation sequencing with a targeted panel.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Yuan, MD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (7):
- China (7):
  - Fujian Medical University Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Affiliated Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - YUANYING, Hangzhou, Zhejinag

IPD SHARING:
Plan to Share IPD: Undecided